CLINICAL TRIAL: NCT03527147
Title: PRISM: A Platform Protocol for the Treatment of Relapsed/Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Platform Study for the Treatment of Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma (PRISM Study)
Acronym: PRISM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-LY-111; 2017-004191-63 (EudraCT Number); D9820C00001 (Other: AstraZeneca); LYM 138 (Other: Sarah Cannon Development Innovations)
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: NHL; DLBCL; Non-hodgkin's Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Acalabrutinib; CALQUENCE®; ACP-196; Platform study; Master protocol; PRISM; Hu-5F9; Rituximab; ATR; STAT3; Anti-CD47; BRD4
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — danvatirsen; acalabrutinib; ceralasertib; magrolimab; Rituximab; AZD5153; MZ1 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD9150 + Acalabrutinib (Experimental): AZD9150 given in combination with acalabrutinib
  Interventions: Drug: AZD9150; Drug: Acalabrutinib
- AZD6738 + Acalabrutinib (Experimental): AZD6738 in combination with acalabrutinib
  Interventions: Drug: Acalabrutinib; Drug: AZD6738
- Hu5F9-G4 + rituximab + Acalabrutinib (Experimental): Hu5F9-G4/rituximab in combination with acalabrutinib
  Interventions: Drug: Acalabrutinib; Drug: Hu5F9-G4; Drug: Rituximab
- AZD5153 + Acalabrutinib (Experimental): AZD5153 in combination with acalabrutinib
  Interventions: Drug: Acalabrutinib; Drug: AZD5153

INTERVENTIONS:
Drug: AZD9150 — AZD9150 will be administered as a 1-hour intravenous (IV) infusion on Days 1, 3, 5 of Cycle 1, followed by weekly infusions (starting Day 8 of Cycle 1 and beyond).
  Other Names: STAT3 inhibitor
  Arms: AZD9150 + Acalabrutinib
Drug: Acalabrutinib — Acalabrutinib will be administered orally twice daily (bid).
  Other Names: CALQUENCE®; ACP-196
Drug: AZD6738 — AZD6738 will be administered orally twice daily (bid).
  Other Names: ATR inhibitor
  Arms: AZD6738 + Acalabrutinib
Drug: Hu5F9-G4 — HU5F9-G4 infusions will be given on Weekly (Day 1, 8, 15, and 22) during the first two 28-day cycles, then will be given every two weeks (Day 1 and Day 15) in Cycle 3 and beyond.
  Other Names: anti-CD47 antibody
  Arms: Hu5F9-G4 + rituximab + Acalabrutinib
Drug: Rituximab — Rituximab infusions will be given Weekly starting on Day 8 (Day 8, 15, and 22) during the first 28-day cycle (4 weeks), then Day 1 of each 4 week cycle for Cycles 2-6. Starting with Cycle 8, Rituximab will be infused on Day 1 of every other cycle (every 8 weeks).
  Other Names: RITUXAN®
  Arms: Hu5F9-G4 + rituximab + Acalabrutinib
Drug: AZD5153 — AZD5153 will be administered orally once per day (qd).
  Other Names: BRD4 inhibitor
  Arms: AZD5153 + Acalabrutinib

SUMMARY:
This is a Phase 1 platform protocol designed to evaluate various targeted agents for the treatment of relapsed/refractory aggressive Non-Hodgkin's Lymphoma (NHL).

DETAILED DESCRIPTION:
This is a Phase 1 platform protocol designed to evaluate various targeted agents for the treatment of relapsed/refractory aggressive Non-Hodgkin's lymphoma (NHL). Each study arm will be conducted in a predefined disease subset. All study arms are open label and allocation to each study arm will not be randomized.

As this master platform protocol has multiple study arms, subjects can be screened for several study arms at once. Likewise, a subject who ends participation in one study arm may be rescreened for participation in another (separate) study arm.

The primary objective of the study is to evaluate the safety of targeted agents for the treatment of relapsed/refractory aggressive Non-Hodgkin's Lymphoma (NHL). This protocol has a modular design, with the potential for future treatment arms to be added via protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria For All Arms:

1. Diagnosis of relapsed/refractory aggressive Non Hodgkin's Lymphoma (NHL) with histology based on established World Health Organization (WHO) criteria.
2. Must have received ≥1 prior line of therapy for the treatment of current histology, there are no known curative treatment options available, or subject ineligible for potential curative options.
3. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy. Not applicable for cutaneous lesions.
4. ECOG performance status of ≤2.

Inclusion Criteria for Arm 1:

1. Must have previously received rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate, and prednisone or equivalent regimen with stem-cell rescue. Or who are ineligible for highdose chemotherapy with stem-cell rescue and/or chimeric antigen receptor (CAR) T cell therapy.

Ineligibility for high-dose therapy with stem cell rescue and/or CAR T-cell therapy will be determined by the investigator.

Inclusion Criteria for Arm 2:

1. Must have previously received rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate, and prednisone or equivalent regimen with stem-cell rescue. Or who are ineligible for highdose chemotherapy with stem-cell rescue and/or chimeric antigen receptor (CAR) T-cell therapy.

Ineligibility for high-dose therapy with stem cell rescue and/or CAR T-cell therapy will be determined by the investigator.

Inclusion Criteria for Arm 3:

1. Must have previously received rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate, and prednisone or equivalent regimen with stem-cell rescue. Or who are ineligible for highdose chemotherapy with stem-cell rescue and/or chimeric antigen receptor (CAR) T cell therapy.

Ineligibility for high-dose therapy with stem cell rescue and/or CAR T-cell therapy will be determined by the investigator.

Inclusion Criteria for Arm 4:

1. Must have previously received rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate, and prednisone or equivalent regimen with stem-cell rescue. Or who are ineligible for highdose chemotherapy with stem-cell rescue and/or chimeric antigen receptor (CAR) T cell therapy.

Ineligibility for high-dose therapy with stem cell rescue and/or CAR T-cell therapy will be determined by the investigator.

Exclusion Criteria:

Exclusion Criteria For All Arms:

1. History of prior malignancy except for the following: a) Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening and felt to be at low risk for recurrence by treating physician, b) Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanomatous skin cancer, c) Adequately treated carcinoma in situ without current evidence of disease, d) Evidence of severe or uncontrolled systemic disease, or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension, history of, or active, bleeding diatheses or uncontrolled active systemic fungal, bacterial, viral, or other infection, or intravenous anti-infective treatment within 2 weeks before first dose of study treatment.
2. Serologic status reflecting active hepatitis B or C infection.
3. Prior use of standard antilymphoma therapy or radiation therapy within 14 days of receiving the first dose of study treatment (not including palliative radiotherapy or palliative corticosteroid use).
4. Requires ongoing immunosuppressive therapy, including systemic corticosteroids for treatment of lymphoid cancer or other conditions.
5. For subjects under DLT review only: Any haematopoietic growth factors or darbepoetin within 14 days of the first dose of study treatment.

Exclusion Criteria for Arm 1:

1. Presence of central nervous system (CNS) lymphoma or leptomeningeal disease.
2. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
3. Requires treatment with proton-pump inhibitors.
4. Requires treatment with strong CYP3A inhibitors or inducers.

Exclusion Criteria for Arm 2:

1. Relative hypotension (< 90/60 mm Hg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of >20 mm Hg.
2. Uncontrolled hypertension requiring clinical intervention.
3. At risk for brain perfusion problems based on medical history.
4. Mean resting QT interval (QTc) calculated using Fridericia's formula (QTcF) >470 msec for female subjects and >450 msec for male subjects obtained from 3 electrocardiograms (ECGs), or congenital long QT syndrome.
5. Presence of central nervous system (CNS) lymphoma or leptomeningeal disease.
6. Known to have tested positive for human immunodeficiency virus (HIV) & requires treatment with restricted medications.
7. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
8. Requires treatment with proton-pump inhibitors.

Exclusion Criteria for Arm 3:

1. Presence of central nervous system (CNS) lymphoma or leptomeningeal disease.
2. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
3. Requires treatment with proton-pump inhibitors.
4. Red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of RBC transfusions during the 4-week period prior to screening.
5. History of haemolytic anaemia or Evans syndrome in the last 3 months before enrolment.
6. Positive IgG component of the direct antiglobulin test (DAT).
7. Prior treatment with CD47 or SIRPα-targeting agents.
8. Hypersensitivity to the active substance or to murine proteins, or to any of the other excipients of rituximab

Exclusion Criteria for Arm 4:

1. Presence of central nervous system (CNS) lymphoma or leptomeningeal disease.
2. Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal (GI) function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
3. Requires treatment with proton-pump inhibitors.
4. Requires treatment with CYP3A inhibitors or inducers or substrates of drug transporters.
5. History of tuberculosis.
6. Mean resting corrected QT interval (QTcF) >450 msec obtained from 3 electrocardiograms (ECGs); clinically important ECG findings, or risk factors for QTc prolongation.
7. Subjects receiving antiplatelet or anticoagulant therapies within 28 days of first dose of study drug.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Safety of the study treatments when given in combination [Incidence of adverse events] | Through to study completion, an average of 1 year
  Incidence of adverse events

SECONDARY OUTCOMES:
Assessment of the efficacy of each treatment by evaluation of overall response rate using RECIL 2017 response criteria | Through to study completion, an average of 1 year
  The overall response rate (ORR) is defined as the rate of subjects who achieve either a partial response (PR) or complete response (CR) as assessed by investigators before receiving any other anticancer therapy.
Duration of response (DOR) using RECIL 2017 response criteria for the anti-tumour activity of each therapy. | Through to study completion, an average of 1 year
  Duration of Response (DOR) is defined as the time from the first objective response of CR or PR to the time of documented disease progression or death due to any cause, whichever occurs first.
Progression free survival (PFS) using RECIL 2017 response criteria for the anti-tumour activity of each therapy. | Through to study completion, an average of 1 year
  Progression free survival (PFS) is defined as the time from first dose date to documented objective disease progression, or death from any cause, whichever occurs first. Disease progression will be determined by the investigators per standard response criteria as outlined in each respective study arm.
Overall Survival (OS) | From the beginning of treatment until the date of death from any cause, assessed up to 12 months
  Overall Survival (OS) is defined as the time from first dose until the date of death from any cause.
Peak plasma concentration (Cmax) of Study Drug A (Arm 1) | Samples will be collected predose and 1, 4, 6 hours postdose on Cycle 1 Day 8 only; then predose and approximately 1 hr (end of infusion of Study Drug A) on Day 1 of every odd cycle starting with Cycle 3 through study completion, an average of 1 year
Peak plasma concentration (Cmax) of Study Drug B (Arm 2) | Samples will be collected predose and 1, 4, 8 hours postdose on Cycle 1 Day 8 only; then predose on Cycle 2 Day 1 and Cycle 3 Day 1
Area under the plasma concentration versus time curve (AUC) of Study Drug A (Arm 1) | Samples will be collected predose and 1, 4, 6 hours postdose on Cycle 1 Day 8 only; then predose and approximately 1 hr (end of infusion of Study Drug A) on Day 1 of every odd cycle starting with Cycle 3 through study completion, an average of 1 year
Area under the plasma concentration versus time curve (AUC) of Study Drug B (Arm 2) | Samples will be collected predose and 1, 4, 8 hours postdose on Cycle 1 Day 8 only; then predose on Cycle 2 Day 1 and Cycle 3 Day 1
Presence of Anti-Drug Antibody (ADA) titres in subjects treated with Study Drug A | Samples will be collected predose on Days 1 and 8 of Cycle 1 and predose on Day 1 of every odd cycle starting with Cycle 3
Peak plasma concentration (Cmax) of acalabrutinib (Arm 1) | Samples will be collected predose and 1, 4, 6 hours postdose on Cycle 1 Day 8 only
Area under the plasma concentration versus time curve (AUC) for acalabrutinib (Arm 1) | Samples will be collected predose and 1, 4, 6 hours postdose on Cycle 1 Day 8 only
Peak plasma concentration (Cmax) of acalabrutinib (Arm 2) | Samples will be collected predose and 1, 4, 8 hours postdose on Cycle 1 Day 8 only; then predose on Cycle 2 Day 1 and Cycle 3 Day 1
Area under the plasma concentration versus time curve (AUC) for acalabrutinib (Arm 2) | Samples will be collected predose and 1, 4, 8 hours postdose on Cycle 1 Day 8 only; then predose on Cycle 2 Day 1 and Cycle 3 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flinn, MD, PhD, Study Chair — Tennessee Oncology
Locations (12):
- United States (10):
  - Research Site, Los Angeles, California
  - Research Site, Sarasota, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, New Orleans, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Omaha, Nebraska
  - Research Site, Rochester, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
- United Kingdom (2):
  - Research Site, London
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-LY-111&attachmentIdentifier=e69332cf-49ef-4d8a-bbd2-1999430907ad&fileName=D9820C00001_CSR_Core+All_Arms_Synopsis_Redacted_Final_Redacted_v2.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search